CLINICAL TRIAL: NCT01388946
Title: Perioperative Ropivacaine Wound Infusion in Laparoscopic Cholecystectomy. A Randomized Controlled Double-blind Trial
Brief Title: Analgesia in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Argyro Fassoulaki, MD, PhD, DEAA, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 149/27.5.10 & Σ-147/03-08-10
Record Dates: First submitted 2011-06-29; First posted 2011-07-07 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Pain, Postoperative; Chronic Postoperative Pain
Keywords: acute postoperative pain; late pain; chronic pain; wound irrigation with local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine 0.75 (Active Comparator): Continuous infusion of ropivacaine 7.5 mg/ml, 2 ml/h for 24 hours
  Interventions: Drug: Ropivacaine 0.75
- Normal saline (Placebo Comparator): Continuous infusion of normal saline 2 ml/h for 24 hours
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine 0.75
  Other Names: Naropeine
  Arms: Ropivacaine 0.75
Drug: Normal saline
  Other Names: 0.9% saline
  Arms: Normal saline

SUMMARY:
The investigators hypothesis is that perioperative infusion of 0.75 ropivacaine in patients undergoing laparoscopic cholecystectomy may modify the intensity of postoperative pain or the analgesic consumption during the first 24 hours.

DETAILED DESCRIPTION:
Patients scheduled for laparoscopic cholecystectomy were randomly assigned to receive via a subcutaneous catheter 2 ml per hour of 0.75 ropivacaine or same volume of normal saline. The catheter was inserted after induction of general anesthesia and before beginning of surgery and continued for the first 24 postoperative hours. The solutions were administered by means of an elastomeric pump. Before induction of anesthesia metoclopramide 10 mg, ranitidine 50 mg and droperidol 0.75 mg were given intravenously. In the operating room the routine monitoring was applied. Anesthesia was induced with thiopental 5-6 mg/kg, fentanyl 2 μg/kg, and rocuronium 0.6 mg/kg, and maintained with sevoflurane 1-1.5 Minimum Alveolar Concentration (MAC) in a nitrous oxide/oxygen mixture. After induction of anesthesia diclofenac 75 mg I.V was given within 30 min. Before wound closure each hole was infiltrated with 2 ml of ropivacaine 0.75 or normal saline. At the end of surgery neuromuscular block was reversed with sugammadex 2 mg/kg., the patient was extubated and transferred to the Post-anesthesia Care Unit (PACU).

Intra-operatively, the intra-abdominal pressure, the rate of carbon dioxide insufflation and the total amount of carbon dioxide insufflated are recorded every 5 minutes.

Besides the ropivacaine infusion in the operative site, postoperative analgesia is assured in the PACU with paracetamol 1 gr and tramadol 100 mg if Visual Analogue Scale (VAS) score is above 40 mm.In the ward Lonarid tablets are given instead.

VAS values and analgesic consumption are recorded in the PACU, and 2, 4, 8, 24 and 48 hours after surgery.

The catheter is removed 24 hours after surgery. One and three months after surgery patients are interviewed by phone for the presence of pain due to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-70 years American Society of Anesthesiology (ASA) physical status I-III
* Scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with chronic pain and/or on analgesics for the last month,
* Patients with central nervous, kidney and liver disease, or allergy to local anesthetics

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Vassi, Principal Investigator — St Savvas Hospital
Locations (2):
- Greece (2):
  - Department of Anesthesia, St Savas Hospital, Athens
  - Aretaieio Hospital, Athens

IPD SHARING:
Plan to Share IPD: No
No plan to share data. The study has been published

RESULTS

PARTICIPANT FLOW:
Groups:
- Ropivacaine 0.75: Continuous infusion of ropivacaine 7.5 mg/ml, 2 ml/h for 24 hours
  Ropivacaine 0.75
- Normal Saline: Continuous infusion of normal saline 2 ml/h for 24 hours
  Normal saline
Period: Overall Study
Arm/Group | Ropivacaine 0.75 | Normal Saline
Started | 55 | 55
Completed | 49 | 52
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Population: To assess differences in patients' characteristics between the two groups, two-independent samples t-tests for normally distributed variables (age and duration of surgery) and Mann-Whitney tests for abnormally distributed variables (BMI and CO2 total volume consumed) were carried out.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.75 | Normal Saline | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 97
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.2) | 48 (12.5) | 50 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  Greece | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: VAS Score Changes ( Cough) During 24 h Postoperatively
Description: Visual Analogue Scale (VAS) measuring pain intensity (mm) with total range 0-100 and with 0 representing no pain and 100 representing possible worst pain.
Time Frame: 24 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary (VAS score at cough) and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 32 (26) | 31 (25)

2. Secondary Outcome: Pain Scores in the Postoperative Care Unit (PACU) at Rest
Description: as for outcome 1
Time Frame: in PACU
Population: Below is the mean and standard deviation of the VAS scores in PACU at rest Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 36 (25) | 46 (21)

3. Secondary Outcome: Pain Scores at Rest 2 h Postoperatively
Description: as for outcome 1
Time Frame: 2 h postoperatively
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery.
  Below are the VAS values (mean and standard deviation) 2 h postoperatively at rest
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 26 (21) | 30 (23)

4. Secondary Outcome: Pain Scores at Rest 4 h Postoperatively
Description: as for outcome 1
Time Frame: 4 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) at rest 4 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 16 (18) | 22 (20)

5. Secondary Outcome: Pain Scores at Rest 8 h Postoperatively
Description: as for outcome 1
Time Frame: 8 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) at rest 8 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 17 (22) | 20 (21)

6. Secondary Outcome: Pain Scores at Rest 24 h Postoperatively
Description: as for outcome 1
Time Frame: 24h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) at rest 24 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 14 (16) | 15 (21)

7. Secondary Outcome: Pain Scores at Rest 48 h Postoperatively
Description: as for outcome 1
Time Frame: 48 h
Population: 50 patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. 1 patient in this group presented ileus after the first 24 h assessment, remaining 49 patients for assessment at 48 hours postoperatively Below are the VAS values (mean and standard deviation) at rest 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 49 | 52
mm | 8 (11) | 12 (15)

8. Secondary Outcome: Pain Scores During Cough in the PACU
Description: as for outcome 1
Time Frame: PACU
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) during cough in PACU
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 42 (27) | 55 (24)

9. Secondary Outcome: Pain Scores During Cough 2 h Postoperatively
Description: as for outcome 1
Time Frame: 2 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) during cough 2 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 36 (27) | 55 (24)

10. Secondary Outcome: Pain Scores During Cough 4 h Postoperatively
Description: as for outcome 1
Time Frame: 4 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) during cough 4 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 25 (19) | 34 (23)

11. Secondary Outcome: Pain Scores During Cough 8 h Postoperatively
Description: as for outcome 1
Time Frame: 8 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) 8 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 50 | 52
mm | 29 (25) | 34 (24)

12. Secondary Outcome: Pain Scores During Cough 48 h Postoperatively
Description: as for outcome 1
Time Frame: 48 h
Population: Fifty patients in the Ropivacaine group were analyzed for the primary and secondary outcomes 24 hours postoperatively. One patient in this group presented ileus after the first 24 h and was not assessed for pain 48 h after surgery Below are the VAS values (mean and standard deviation) during cough 48 h postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 49 | 52
mm | 18 (17) | 26 (21)

13. Secondary Outcome: Chronic Pain
Description: Number and incidence of patients with persisting pain (burning pain, loss of sensation) one month postoperatively
Time Frame: one month postoperatively
Population: Below the number of patients with pain one month postoperatively For the chronic pain assessment in the control group we had two dropouts as contact for two patients was not feasible.
Measure: Number; unit: number of participants
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 49 | 50
number of participants | 5 | 7

14. Secondary Outcome: Chronic Pain
Description: Number and incidence of patients with persisting pain (burning pain, loss of sensation) three month postoperatively
Time Frame: three months
Population: Below the number of patients with pain three months postoperatively. For the chronic pain assessment in the control group we had two dropouts as contact for two patients was not feasible.
Measure: Number; unit: Number of participants
Arm/Group | Ropivacaine 0.75 | Normal Saline
Number analyzed (Participants) | 49 | 50
Number of participants | 2 | 4

ADVERSE EVENTS:
Time Frame: According to study design no adverse events were planned to be collected but in case of adverse events these are routinely included in patient's records for 24 hours postoperatively
Arm/Group | Ropivacaine 0.75 | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No